CLINICAL TRIAL: NCT01442038
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Effects of Ranolazine on Major Adverse Cardiovascular Events in Subjects With a History of Chronic Angina Who Undergo Percutaneous Coronary Intervention With Incomplete Revascularization
Brief Title: Ranolazine for Incomplete Vessel Revascularization Post-Percutaneous Coronary Intervention (PCI)
Acronym: RIVER-PCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-259-0116; 2011-002507-15 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Artery Disease; Angina Pectoris
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Experimental)
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Subjects will receive ranolazine 500 milligrams (mg) twice daily for 7 days, followed by 1000 mg administered orally twice daily for the duration of the study.
  Subjects receiving a moderate CYP3A4 inhibitor will receive ranolazine 500 mg or placebo administered orally twice a day for the duration of the concomitant therapy.
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Subjects will receive one tablet of matching placebo twice daily for 7 days, followed by two tablets of matching placebo twice daily for the duration of the study.
  Subjects receiving a moderate CYP3A4 inhibitor will receive ranolazine 500 mg or placebo administered orally twice a day for the duration of the concomitant therapy.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of ranolazine as compared with placebo when used as part of standard medical therapy in chronic angina subjects with incomplete revascularization post-percutaneous coronary intervention (PCI; formerly known as angioplasty with stent) on the composite of ischemia-driven revascularization or ischemia-driven hospitalization without revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Males and females aged 18 years and older
3. History of chronic angina defined as at least 2 episodes of anginal pain or discomfort in the chest, jaw, shoulder, back, neck, or arm that is precipitated by exertion or emotional stress, and relieved by rest or sublingual nitroglycerin, which occurred on at least 2 separate days and at least 14 days prior to PCI (in the case of staged PCI procedures, at least 14 days prior to the first PCI in the series). Participants may or may not have additional angina episodes within the 14 days prior to their first PCI in the series, as well as any time prior to Randomization.
4. PCI for any indication (ACS or non-ACS). For the purposes of stratification at randomization, ACS will be defined as hospitalization for anginal pain or discomfort within the previous 24 hours to their hospitalization with any one (or more) of the following criteria:

   i. Elevated troponin or creatinine kinase-MB (CK-MB) consistent with myocardial infarction (MI), as reported by local laboratory and measured prior to index PCI ii. Electrocardiographic changes (including transient changes) comprising new or presumably new ST segment depression ≥ 0.1 mV (≥ 1 mm), or ST segment elevation ≥ 0.1 mV (≥ 1 mm) in at least 2 contiguous leads, or new or presumably new Left Bundle Branch Block
5. Randomization within 14 days post-PCI. In the case of staged PCI procedures, randomization has to occur within 14 days of the last PCI in the series. Participants may be randomized starting on the day of PCI and anytime during the following 14 days. PCI is defined as an attempt to cross the lesion with a wire with the intention of performing revascularization.
6. Post-PCI (post the last PCI for staged procedures) evidence of incomplete revascularization defined as the presence of one or more visually estimated ≥ 50% stenoses in one or more coronary arteries with reference vessel diameter of at least 2.0 mm, whether in the target vessel or in a non-target vessel regardless of the presence or absence of coronary collaterals. In the case of a participant post-coronary artery bypass grafting (CABG), incomplete revascularization is defined as the presence of one or more visually estimated ≥ 50% stenoses in an unbypassed epicardial vessel with a reference diameter of ≥ 2.0 mm, or one or more visually estimated ≥ 50% stenoses in a bypass graft supplying an otherwise unrevascularized myocardial territory.
7. Clinically stable post-PCI. Participants randomized in-hospital on day of planned discharge or in clinic are considered stable. Participants randomized in-hospital prior to day of planned discharge must meet all of the following criteria:

   i. CK-MB < 3 times the upper limit of normal (ULN) at least 3 hours post-PCI, or if ≥ 3 times the ULN with evidence of decreasing CK-MB (decreased by at least 20% from the prior measurement) as reported by local laboratory. If CK-MB is not available, a participant must have evidence of normal or decreasing troponin levels (by at least 20% from the prior measurement) at least 3 hours post-PCI, as reported by local laboratory.

   ii. Systolic blood pressure ≥ 90 mm Hg and not receiving pressors or inotropes iii. No current requirement for an intra-aortic balloon pump (IABP) or any left ventricular assist device iv. No current requirement for intravenous (IV) nitroglycerin
8. Ability and willingness to comply with all study procedures during the course of the study
9. Females of childbearing potential must have a negative pregnancy test at Screening (unless surgically sterile or post-menopausal) and must agree to use highly effective contraception methods from Screening throughout the duration of study treatment and for 14 days following the last dose of study drug.

Exclusion Criteria:

1. Any future planned revascularization (including staged procedures) or possible planned revascularization (ie, planned stress test to assess the imminent need for additional revascularization). Future planned stress tests for purposes of monitoring are permitted but strongly discouraged. Participants may be enrolled after the last PCI in the staged series or once a decision is made not to perform a follow up PCI, as long as Randomization occurs within 14 days from the last PCI. If a participant has had a stress test post-PCI and prior to Randomization and no further intervention is planned, the participant may be enrolled within 14 days from the last PCI.
2. Unrevascularized left main coronary artery stenosis ≥ 50%. Participants with a history of CABG to the left coronary system will be considered to have a revascularized left main if at least one graft is patent.
3. Major complication during or after the index PCI (in the case of staged PCI, the last in the series) including:

   i. Major bleeding (TIMI Bleeding classification or any bleeding requiring blood transfusion of ≥ 2 units of red blood cells) ii. Coronary perforation requiring treatment iii. Procedural complication requiring surgery (including CABG or peripheral vascular surgery)
4. Stroke within 90 days prior to Randomization, or any history of stroke with permanent major neurologic disability (eg, aphasia or significant motor dysfunction)
5. Cardiogenic shock within 90 days prior to Randomization (transient decreases in blood pressure without clinical sequelae are not considered to be cardiogenic shock)
6. New York Heart Association (NYHA) Class III or IV heart failure
7. Severe renal insufficiency as assessed by an estimated glomerular filtration rate < 30 mL/min/1.73m2 using the 4 variable modification of diet in renal disease (MDRD) equation per local laboratory (based on the last available measurement prior to Randomization, collected within 1 month prior to the index PCI [in the case of staged PCI, the last in the series])
8. Liver cirrhosis
9. Use of Class Ia, Ic, or Class III antiarrhythmics, except for amiodarone
10. Current treatment with strong inhibitors of CYP3A
11. Current treatment with CYP3A4 inducers or P-gp inducers
12. Participants taking > 20 mg simvastatin daily or > 40 mg lovastatin daily who cannot reduce the dose to 20 mg once daily for simvastatin or 40 mg once daily for lovastatin, or who cannot switch to another statin
13. Participants taking greater than a total of 1000 mg daily of metformin who cannot reduce the dose to a maximum total of 1000 mg daily (additional anti-diabetic medications may be added as clinically indicated to allow participants to decrease their metformin dose and maintain glycemic control)
14. Previous treatment with ranolazine for > 7 consecutive days within 30 days prior to Randomization, or known hypersensitivity or intolerance to ranolazine or to any of the excipients
15. Participation in another investigational drug or investigational device study within 30 days prior to Randomization (participation in registries is allowed)
16. Women who are pregnant or breast feeding
17. Non-coronary artery disease comorbid conditions (eg, advanced malignancy, severe aortic stenosis) which are likely to result in death within 2 years of Randomization
18. Any condition that in the opinion of the investigator would preclude compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2651 (Actual)
Dates: Start 2011-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian McNabb, MD, Study Director — Gilead Sciences
Locations (217):
- United States (85):
  - Cardiology, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - Spectrum Clinical Research Institute, Inc, Moreno Valley, California
  - Veterans Affairs San Diego Healthcare System, San Diego, California
  - John Muir Medical Center Concord Campus, Walnut Creek, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Cardiology Associates of Fairfield County, PC, Stamford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Zasa Clinical Research, Atlantis, Florida
  - Cardiology Research Associates, Daytona Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Michigan Heart, PC, Hialeah, Florida
  - Jacksonville Heart Center, Jacksonville, Florida
  - University of Florida Health Sciences Center-Jacksonville, Jacksonville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Heart Institute, Orlando, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Pepin Heart Hospital and Dr. Kiran C. Patel Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Gateway Cardiology, PC, Jerseyville, Illinois
  - Indiana Heart Physicians, Inc., Indianapolis, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Northwest Indiana Cardiovascular Physicians, Valparaiso, Indiana
  - Iowa Heart Center, West de Moines, Iowa
  - Saint Joseph Cardiology Associates, Lexington, Kentucky
  - Clinical Trials of America, Inc., Minden, Louisiana
  - Clinical Trials of America, Inc., Shreveport, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - Baltimore Heart Associates, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Saint Elizabeth's Medical Center, Boston, Massachusetts
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Essentia Health, Duluth, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Saint John's Regional Medical Center, Springfield, Missouri
  - Gateway Cardiology, PC, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Buffalo Heart Group, Buffalo, New York
  - SJH Cardiology Associates, Liverpool, New York
  - Columbia University Medical Center, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Central New York Cardiology, Utica, New York
  - Westchester Medical Center, Valhalla, New York
  - Buffalo Cardiology and Pulmonary Associates, PC, Williamsville, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Veterans Affairs Medical Center, Duke University Medical Center, Durham, North Carolina
  - Carolina Cardiology Associates, High Point, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - Cardiology Associates of Southeast Ohio, Inc., Zanesville, Ohio
  - Oklahoma City Veterans' Affairs Medical Center, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - The Heart and Vascular Center, Beaver, Pennsylvania
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Saint Vincent Health Care Center, Erie, Pennsylvania
  - Veterans Administration Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health System, Wormleysburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Research Associates of Jackson, Jackson, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Centennial Heart Cardiovascular Consultants, LLC, Nashville, Tennessee
  - North Texas Healthcare System, Dept. of Veteran's Affairs, Dallas, Texas
  - Humble Cardiology Associates, Humble, Texas
  - Gamma Medical Research Inc., Mission, Texas
  - San Antonio Endovascular and Heart Institute, San Antonio, Texas
  - Victoria Heart and Vascular Center, Victoria, Texas
  - Utah Cardiology, PC, Layton, Utah
  - University of Vermont Medical Center, Fletcher Allen Health Care, Burlington, Vermont
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
- Austria (6):
  - Landesklinikum Sankt Pölten, Sankt Pölten, Lower Austria
  - Landeskrankenhaus Graz West, Graz, Styria
  - Innsbruck Universitaetsklinik, Innsbruck, Tyrol
  - Allgemeines Krankenhaus der Stadt Linz, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna, Vienna
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp, Antwerpen
  - Imelda Ziekenhuis, Bonheiden, Antwerpen
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège, Liege
  - ZOL Genk, Campus Saint Jan, Genk, Limburg
  - Algemeen Ziekenhuis Sint-Jan, Bruges, West-Vlaanderen
- Canada (13):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - Hamilton Health Sciences, General Site, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Scarborough Cardiology Research Associates, Scarborough Village, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Czechia (8):
  - Karlovarská krajská nemocnice a.s., Karlovy Vary, Karlovarský kraj
  - Krajská nemocnice Liberec a.s., Liberec, Liberecký kraj
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice u sv. Anny v Brne, Brno
  - Fakultní nemocnice Olomouc, Olomoucký Kraj
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Fakultní Nemocnice v Motole, Prague
- France (5):
  - Centre Hospitalier d'Annecy, Pringy, Auvergne-Rhône-Alpes
  - Centre Hospitalier d'Arras, Arras, Hauts-de-France
  - Hôpital Rangueil, Toulouse, Midi-Pyrenees
  - Groupe hospitalier La Pitié Salpêtrière, Paris
  - Hôpital Bichat-Claude Bernard, Paris, Île-de-France Region
- Germany (8):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Kerckhoff-Klinik GmbH, Bad Nauheim, Hesse
  - Asklepios-Kliniken Langen, Langen, Hesse
  - Städtische Kliniken Bielefeld gGmbH, Bielefeld, North Rhine-Westphalia
  - Sankt Johannes Hospital, Dortmund, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Krankenhaus Der Barmherzigen Brüder Trier, Trier, Rhineland-Palatinate
  - Vivantes Klinikum im Friedrichshain, Berlin, State of Berlin
- Israel (15):
  - Kaplan Medical Center, Rehovot, Reheoboth
  - HaEmek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Assaf Harofeh Medical Centre, Beer Yahkov
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein-Kerem Medical Centre, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital, Nahariya
  - Hillel Yaffe Medical Center, Ramat Gan
  - Tel Aviv Souraski Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - ZIV Medical Center, Zafed
- Italy (9):
  - Ospedali Riuniti di Bergamo, Bergamo, Bergamo
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Firenze
  - Azienda Ospedaliera Universitaria San Martino, Genova, Genova
  - Fondazione Centro S. Raffaele del Monte Tabor, Ospedale San Raffaele, Milan, Milano
  - Ospedale Civile SS Annunziata ASL 1, Sassari, Sassari
  - Azienda Ospedaliera S. Sebastiano di Caserta, Caserta
  - Azienda Ospedaliera "Maggiore della Carita" di Novara, Novara
  - A.R.N.A.S. Civico G. Di Cristina Benfratelli, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
- Netherlands (5):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Ziekenhuis Rijnstate Arnhem, Gelderland
- Poland (17):
  - American Heart of Poland S.A., Chrzanów, Lesser Poland Voivodeship
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - 4th Wojskowy Szpital Kliniczny z Poliklinika, Klinika Kardiologii, Wroclaw, Lower Silesian Voivodeship
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw, Masovian Voivodeship
  - Instytut Kardiologii, Warsaw, Masovian Voivodeship
  - American Heart of Poland S.A., Kędzierzyn-Koźle, Opole Voivodeship
  - American Heart of Poland S.A., Mielec, Podkarpackie Voivodeship
  - American Heart of Poland S.A., Bielsko-Biala, Silesian Voivodeship
  - American Heart of Poland S.A., Dabrowa Górnicza, Silesian Voivodeship
  - SPZOZ, SPSK nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach, Górnoslaskie Centrum Medyczne, Katowice, Silesian Voivodeship
  - American Heart of Poland S.A., Tychy, Silesian Voivodeship
  - American Heart of Poland S.A., Ustroń, Silesian Voivodeship
  - SPZOZ, Szpital Wojewódzki we Wloclawku, Kujawsko-pomorskie
  - Samodzielny Publiczny Szpital Kliniczny nr. 1 im. Przemienienia Panskiego, Poznan
  - Wojewódzki Szpital Zespolony im. Ludwika Rydygiera w Toruniu, Torun
  - SPZOZ, Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw
  - American Heart of Poland S.A., Belchatów, Łódź Voivodeship
- Russia (19):
  - Altai Regional Cardiological Dispensary, Barnaul
  - Regional Clinical Hospital №3, Chelyabinsk
  - Cardiological Dispensary, Ivanovo
  - Republic Clinical Hospital № 2, Kazan'
  - Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo
  - Medical Center "Alliance", Kirovsk, Leningradskaya Region
  - Regional Clinical Hospital, Krasnoyarsk
  - National Research Center For Preventive Medicine, Moscow
  - City Clinical Hospital # 23 n.a."Medsantrud", Moscow
  - City Clinical Hospital #15 named after O.M. Filatov, Moscow
  - University Clinical Hospital #1, Moscow
  - City Clinical Hospital n.a. S.P.Botkin, Moscow
  - City Clinical Hospital #5, Nizhny Novgorod
  - City Clinical Emergency Hospital # 2, Novosibirsk
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - Federal Center of Heart, Blood and Endocrinology n.a. V.A.Almazov, Saint Petersburg
  - Scientific and Research Institution Of Cardiology, Tomsk
  - Volgograd Regional Clinical Cardiological Center, Volgograd
  - Ural Institute of Cardiology, Yekaterinburg
- Spain (11):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Vall d´Hebrón, Barcelona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Complejo Hospitalario Universitario de Vigo, Meixoeiro Hospital, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (5):
  - Uppsala University Hospital, Uppsala, Uppsala County
  - Falu lasarett, Falun
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Karlstad Central Hospital, Karlstad
  - Universitetssjukhuset Örebro, Örebro, Örebro County
- United Kingdom (6):
  - Royal Sussex County Hospital, Brighton, England
  - The James Cook University Hospital, Middlesbrough, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Ashford and Saint Peter's Hospital NHS Trust, Surrey, England
  - Saint Richards Hospital, West Sussex, England
  - Royal Victoria Hospital, Northern Ireland

REFERENCES:
- [Background] Weisz G, Farzaneh-Far R, Ben-Yehuda O, Debruyne B, Montalescot G, Lerman A, Mahmud E, Alexander KP, Ohman EM, White HD, Olmsted A, Walker GA, Stone GW. Use of ranolazine in patients with incomplete revascularization after percutaneous coronary intervention: design and rationale of the Ranolazine for Incomplete Vessel Revascularization Post-Percutaneous Coronary Intervention (RIVER-PCI) trial. Am Heart J. 2013 Dec;166(6):953-959.e3. doi: 10.1016/j.ahj.2013.08.004. Epub 2013 Oct 16. PMID 24268208
- [Result] Weisz G, Genereux P, Iniguez A, Zurakowski A, Shechter M, Alexander KP, Dressler O, Osmukhina A, James S, Ohman EM, Ben-Yehuda O, Farzaneh-Far R, Stone GW; RIVER-PCI investigators. Ranolazine in patients with incomplete revascularisation after percutaneous coronary intervention (RIVER-PCI): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2016 Jan 9;387(10014):136-45. doi: 10.1016/S0140-6736(15)00459-6. Epub 2015 Oct 22. PMID 26474810
- [Result] Alexander KP, Weisz G, Prather K, James S, Mark DB, Anstrom KJ, Davidson-Ray L, Witkowski A, Mulkay AJ, Osmukhina A, Farzaneh-Far R, Ben-Yehuda O, Stone GW, Ohman EM. Effects of Ranolazine on Angina and Quality of Life After Percutaneous Coronary Intervention With Incomplete Revascularization: Results From the Ranolazine for Incomplete Vessel Revascularization (RIVER-PCI) Trial. Circulation. 2016 Jan 5;133(1):39-47. doi: 10.1161/CIRCULATIONAHA.115.019768. Epub 2015 Nov 10. PMID 26555329
- [Derived] Fanaroff AC, Prather K, Brucker A, Wojdyla D, Davidson-Ray L, Mark DB, Williams RB, Barefoot J, Weisz G, Ben-Yehuda O, Stone GW, Ohman EM, Alexander KP. Relationship Between Optimism and Outcomes in Patients With Chronic Angina Pectoris. Am J Cardiol. 2019 May 1;123(9):1399-1405. doi: 10.1016/j.amjcard.2019.01.036. Epub 2019 Feb 7. PMID 30771861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Canada, Europe, Russia, and Israel. The first participant was screened on 03 November 2011. The last study visit occurred on 09 February 2015.
Pre-assignment Details: 2734 participants were screened.
Groups:
- Ranolazine: Ranolazine 500 mg (1 x 500 mg tablet) twice daily for 7 days, followed by ranolazine 1000 mg (2 x 500 mg tablet) twice daily for the duration of the study (participants receiving a moderate CYP3A4 inhibitor continued to receive ranolazine 500 mg (1 x 500 mg tablet) twice daily for the duration of the study)
- Placebo: Ranolazine placebo (1 tablet) for 7 days, followed by ranolazine placebo (2 tablets) twice daily for the duration of the study (participants receiving a moderate CYP3A4 inhibitor continued to receive ranolazine placebo (1 tablet) twice daily for the duration of the study)
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 1332 | 1319
Completed | 1029 | 1040
Not Completed | 303 | 279
Not completed — Death | 35 | 29
Not completed — Investigator-Initiated Early Closure | 44 | 43
Not completed — Participant Withdrew Consent | 137 | 102
Not completed — Lost to Follow-up | 37 | 51
Not completed — Adverse Event | 26 | 15
Not completed — Protocol Deviation | 9 | 20
Not completed — Investigator's Discretion | 13 | 16
Not completed — Study Terminated By Sponsor | 2 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participant who were randomized and received at least one dose of study drug
Groups:
- Placebo: Ranolazine placebo (1 tablet) twice daily for 7 days, followed by ranolazine placebo (2 tablets) twice daily for the duration of the study (participants receiving a moderate CYP3A4 inhibitor continued to receive ranolazine placebo (1 tablet) twice daily for the duration of the study)
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 1322 | 1297 | 2619
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.51) | 63.4 (10.06) | 63.4 (10.29)
Age, Customized [Number; unit: participants]
  < 65 Years | 714 | 719 | 1433
  65-74 Years | 402 | 383 | 785
  ≥ 75 Years | 206 | 195 | 401
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 260 | 536
  Male | 1046 | 1037 | 2083
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 16 | 10 | 26
  Black or African American | 49 | 43 | 92
  Native Hawaiian or Pacific Islander | 2 | 1 | 3
  White | 1203 | 1196 | 2399
  Other | 29 | 28 | 57
  Not Permitted | 23 | 16 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 72 | 64 | 136
  Not Hispanic or Latino | 1219 | 1208 | 2427
  Not Reported | 28 | 24 | 52
  Unknown | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Russian Federation | 154 | 168 | 322
  United States | 499 | 466 | 965
  United Kingdom | 16 | 17 | 33
  Spain | 80 | 87 | 167
  Canada | 80 | 85 | 165
  Austria | 12 | 15 | 27
  Czech Republic | 31 | 44 | 75
  Netherlands | 13 | 13 | 26
  Sweden | 19 | 25 | 44
  Belgium | 20 | 21 | 41
  Poland | 203 | 172 | 375
  Italy | 28 | 33 | 61
  Israel | 111 | 109 | 220
  France | 22 | 15 | 37
  Germany | 34 | 27 | 61

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates for Time From Randomization to First Occurrence of Ischemia-driven Revascularization or Ischemia-driven Hospitalization Without Revascularization
Description: Time to event distributions were estimated by the Kaplan-Meier (KM) method. 1 month = 28 days; 1 calendar year = 365 days.
Time Frame: Baseline through end of study (average 90 weeks)
Population: Full Analysis Set: all participants in the Safety Analysis Set (randomized and received at least one dose of study drug), except participants with no qualifying percutaneous coronary intervention (PCI; formerly known as angioplasty with stent))
Measure: Number; unit: percentage of participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 1317 | 1287
percentage of participants
  KM Estimate: 1 Month | 3.4 | 2.3
  KM Estimate: 6 Months | 11.3 | 10.0
  KM Estimate: 12 Months | 19.1 | 17.3
  KM Estimate: 1 Calendar Year | 20.2 | 18.9
  KM Estimate: 18 Months | 23.8 | 25.3
  KM Estimate: 24 Months | 27.6 | 29.4
  KM Estimate: 2 Calendar Years | 30.7 | 31.0
  KM Estimate: 30 months | 31.1 | 33.8
  KM Estimate: 36 Months | 32.2 | 37.8
  KM Estimate: 3 Calendar Years | NA — NA = not calculable: all participants had an event or were censored prior to the Year 3 time point | 37.8
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.48, Cox Proportional Hazards Model — The p-value and hazard ratio are from Cox proportional hazards model stratifying by reason for qualifying percutaneous coronary intervention (PCI): acute coronary syndrome (ACS) versus non-ACS indication, and history of diabetes (yes versus no); Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.818 to 1.099]

2. Secondary Outcome: Kaplan-Meier Estimates for Time From Randomization to Sudden Cardiac Death
Description: Time to event distributions were estimated by the Kaplan-Meier method. 1 month = 28 days; 1 calendar year = 365 days.
Time Frame: Baseline through end of study (average 90 weeks)
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 1317 | 1287
percentage of participants
  KM Estimate: 1 Month | 0.2 | 0.1
  KM Estimate: 6 Months | 0.5 | 0.2
  KM Estimate: 12 Months | 0.5 | 0.5
  KM Estimate: 1 Calendar Year | 0.5 | 0.5
  KM Estimate: 18 Months | 0.5 | 0.8
  KM Estimate: 24 Months | 0.5 | 0.9
  KM Estimate: 2 Calendar Years | 0.7 | 0.9
  KM Estimate: 30 months | 0.7 | 0.9
  KM Estimate: 36 Months | 0.7 | 0.9
  KM Estimate: 3 Calendar Years | 0.7 | 0.9
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.40, Cox Proportional Hazards Model — The p-value and hazard ratio are from Cox proportional hazards model stratifying by reason for qualifying PCI: ACS versus non-ACS indication, and history of diabetes (yes versus no); Hazard Ratio (HR) = 0.665, 95% CI 2-sided [0.244 to 1.691]

3. Secondary Outcome: Kaplan-Meier Estimates for Time From Randomization to Cardiovascular Death
Description: Time to event distributions were estimated by the Kaplan-Meier method. 1 month = 28 days; 1 calendar year = 365 days.
Time Frame: Baseline through end of study (average 90 weeks)
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 1317 | 1287
percentage of participants
  KM Estimate: 1 Month | 0.2 | 0.1
  KM Estimate: 6 Months | 0.6 | 0.4
  KM Estimate: 12 Months | 1.0 | 0.9
  KM Estimate: 1 Calendar Year | 1.1 | 1.0
  KM Estimate: 18 Months | 1.5 | 1.4
  KM Estimate: 24 Months | 1.7 | 1.7
  KM Estimate: 2 Calendar Years | 1.9 | 1.7
  KM Estimate: 30 months | 1.9 | 1.7
  KM Estimate: 36 Months | 1.9 | 1.7
  KM Estimate: 3 Calendar Years | 1.9 | 1.7
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.82, Cox Proportional Hazards Model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.579 to 1.994]

4. Secondary Outcome: Kaplan-Meier Estimates for Time From Randomization to Myocardial Infarction
Description: Time to event distributions were estimated by the Kaplan-Meier method. 1 month = 28 days; 1 calendar year = 365 days.
Time Frame: Baseline through end of study (average 90 weeks)
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 1317 | 1287
percentage of participants
  KM Estimate: 1 Month | 1.2 | 0.6
  KM Estimate: 6 Months | 3.8 | 3.3
  KM Estimate: 12 Months | 5.8 | 5.7
  KM Estimate: 1 Calendar Year | 6.2 | 6.2
  KM Estimate: 18 Months | 7.3 | 8.5
  KM Estimate: 24 Months | 8.7 | 9.4
  KM Estimate: 2 Calendar Years | 10.0 | 9.4
  KM Estimate: 30 months | 10.9 | 10.1
  KM Estimate: 36 Months | 10.9 | 13.4
  KM Estimate: 3 Calendar Years | 10.9 | 13.4
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.81, Cox Proportional Hazards Model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.745 to 1.256]

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure 72 weeks) plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 516/1322 | 485/1297
Other Adverse Events (participants affected / at risk) | 665/1322 | 531/1297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=1322) | Placebo (N=1297)
Anaemia (Blood and lymphatic system disorders) | 10 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Platelet dysfunction (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 9
Acute myocardial infarction (Cardiac disorders) | 28 | 29
Angina pectoris (Cardiac disorders) | 125 | 114
Angina unstable (Cardiac disorders) | 58 | 71
Arrhythmia (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 12 | 14
Atrial flutter (Cardiac disorders) | 5 | 0
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 5 | 3
Cardiac arrest (Cardiac disorders) | 5 | 3
Cardiac failure (Cardiac disorders) | 11 | 12
Cardiac failure acute (Cardiac disorders) | 2 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 20 | 6
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 14 | 11
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 4
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 18 | 18
Myocardial ischaemia (Cardiac disorders) | 8 | 12
Myocardial rupture (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 2
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 2
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 5 | 4
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Hyphaema (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2
Duodenitis (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 13
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Radicular cyst (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 6 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 3
Arterial restenosis (General disorders) | 0 | 2
Asthenia (General disorders) | 3 | 0
Carotid artery restenosis (General disorders) | 1 | 0
Chest discomfort (General disorders) | 2 | 3
Chest pain (General disorders) | 37 | 24
Coronary artery restenosis (General disorders) | 1 | 2
Death (General disorders) | 1 | 1
Device extrusion (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Impaired healing (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 19 | 19
Oedema peripheral (General disorders) | 0 | 1
Peripheral artery restenosis (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 2
Sudden cardiac death (General disorders) | 2 | 1
Thrombosis in device (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 2 | 1
Abscess neck (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 3
Appendicitis perforated (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 4
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Bursitis infective (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 5 | 2
Cholangitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 4 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Gingival abscess (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 1
Osteomyelitis acute (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 14 | 12
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 3
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 6
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Cardiac stress test abnormal (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 1 | 0
Carotid artery dissection (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 8 | 2
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 12 | 9
Dizziness (Nervous system disorders) | 5 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 5 | 1
Lacunar infarction (Nervous system disorders) | 0 | 2
Lateral medullary syndrome (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Mononeuropathy (Nervous system disorders) | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 9 | 2
Radicular pain (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 25 | 13
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 12 | 3
Tremor (Nervous system disorders) | 1 | 0
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 4
Suicidal ideation (Psychiatric disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 4
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 0
Renal failure acute (Renal and urinary disorders) | 5 | 6
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 4
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 5 | 2
Aortic stenosis (Vascular disorders) | 3 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 9 | 3
Hypertensive crisis (Vascular disorders) | 1 | 2
Hypertensive emergency (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 7 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 3 | 0
Ischaemia (Vascular disorders) | 0 | 1
Lymphorrhoea (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 4 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 7
Peripheral artery stenosis (Vascular disorders) | 1 | 2
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 6 | 7
Peripheral vascular disorder (Vascular disorders) | 4 | 5
Renovascular hypertension (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=1322) | Placebo (N=1297)
Angina pectoris (Cardiac disorders) | 161 | 156
Constipation (Gastrointestinal disorders) | 167 | 71
Nausea (Gastrointestinal disorders) | 123 | 63
Chest pain (General disorders) | 97 | 92
Fatigue (General disorders) | 99 | 74
Dizziness (Nervous system disorders) | 240 | 119
Headache (Nervous system disorders) | 98 | 89
Cough (Respiratory, thoracic and mediastinal disorders) | 69 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 89 | 89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years